CLINICAL TRIAL: NCT01151514
Title: Referral Patterns for Hospital Acquired Acute Kidney Injury and Relevance to Renal Outcomes
Acronym: HA-AKI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Other Study IDs: HA-AKI referral
Record Dates: First submitted 2010-06-23; First posted 2010-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-08

CONDITIONS: Renal Replacement Therapy; Mortality
Keywords: No referral; Late referral; Acute kidney injury; Intensive care unit; In-hospital mortality; Renal outcome; Requirement for renal replacement therapy; Length of hospital stay; Impact; Incidence
MeSH Terms: conditions — Acute Kidney Injury; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- nrHA-AKI patients: Patients with hospital-acquired acute kidney injury not referred to the nephrologists
  Interventions: Other: Nephrologist referral
- lrHA-AKI patients: Patients with hospital-acquired acute kidney injury whao are late referred to the nephrologists
  Interventions: Other: Nephrologist referral

INTERVENTIONS:
Other: Nephrologist referral — Nephrologist specialty, renal replacement therapy
  Other Names: Control group: early-referred patients with HA-AKI.

SUMMARY:
Few studies analyzed the referral time to nephrologists and its impact on the patient outcome in a large cohort. The investigators described the incidence and determined the outcome with respect to renal function recovery, renal replacement therapy (RRT) requirement and in-hospital mortality of Hospital Acquired Acute Kidney Injury (HA-AKI) without nephrology referral (nrHA-AKI) and late referred HA-AKI patients to nephrologists (lrHA-AKI) compared with early referral patients (erHA-AKI). The patients included were admitted to the tertiary care academic center of Lausanne (Switzerland) between 2004 and 2008, in the medical and surgical services and in the intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* Hospitalization in the medicine and surgery wards and in the intensive care unit.
* Hospitalized patients with acquired acute kidney injury according to the
* Acute Kidney Injury Network (AKIN)criteria.
* HA-AKI patients with no referral to the nephrologist (nrHA-AKI).
* HA-AKI patients referred late (more than five days [> 5 days]) to the nephrologist (lrHA-AKI).
* HA-AKI patients early referred (within five days after sCr increase) to the nephrologist (erHA-AKI).

Exclusion Criteria:

* Patients with AKI at the time of the hospital admission and during the first
* 48 hours after admission.
* Patients hospitalized in other wards.
* Children under 18.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population consisted of patients who were hospitalized in the medical and surgical departments as well as in the intensive care untis (ICU) of the University Hospital of Lausanne (Centre Hospitalier Universitaire Vaudois [CHUV]) that is a tertiary care academic medical center. Patients with AKI coming from ICU in the medicine or surgery wards, and patients from medicine or surgery wards, who required a transfer to ICU during the hospital stay, were also included whatever the cause of the transfer.
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
Referral patterns for hospital acquired acute kidney injury and relevance to renal outcomes
  Recovery of renal function during hospital stay. Requirement for renal replacement therapy.

SECONDARY OUTCOMES:
Referral patterns for hospital acquired acute kidney injury and relevance to renal outcomes
  Length of hospital stay. In-hospital mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology - CHCVs, Sion, Switzerland

REFERENCES:
- See also: Related Info — http://www.chuv.ch